CLINICAL TRIAL: NCT04777045
Title: Efficacy of Diltiazem to Improve Coronary Microvascular Dysfunction: a Randomized Clinical Trial
Acronym: EDIT-CMD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL67497.091.19; 2018-003518-41 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-03-02 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-10

CONDITIONS: Microvascular Angina; Coronary Vasospasm; Microvascular Ischemia of Myocardium
Keywords: Coronary vasospasm; IMR; CFR; Diltiazem; Coronary function testing
MeSH Terms: conditions — Microvascular Angina; Coronary Vasospasm | interventions — Diltiazem

STUDY DESIGN:
Intervention Model Description: A clinical multi-center randomized with 1:1 ratio, double-blind, placebo-controlled study. Patients with chronic angina in the absence of CAD will be screened for study enrolment. Eligible patients will be asked for informed consent at the screening visit.
  Within 8 weeks after screening, participants undergo coronary function testing. If this shows either a CFR ≤ 2.0, an IMR ≥ 25 and/or abnormal acetylcholine testing the patient will continue in the intervention arm and will be randomized to either diltiazem or placebo treatment for 6 weeks. After 6 weeks, coronary function testing will be repeated and the diltiazem/placebo treatment will be discontinued. Follow-up will be obtained 1 month, 1 year and 5 years after treatment discontinuation. If coronary function testing at baseline shows no signs of vascular dysfunction, patients will enter in the registration arm of the study. These patients will not receive any study medication. Follow-up will be obtained after 1 year and 5 years.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinding of treatment is ensured by using a double-blind technique. The diltiazem capsules and the respective placebo capsules will have the same look and feel. The bottles with the IMP will be labelled with unique identification numbers. No member of the study team, or anyone handling study data will have access to the randomization scheme during the study. In case of an adverse event (AE), the code should only be broken in circumstances when knowledge of the IMP is required for treating the patient. If possible, contact should be initiated with the principal investigator before breaking the code. Code breaking can be performed at any time by the investigator. A sealed emergency envelope per patient randomization number will be present per patient at the research department. If the blind is broken, the Investigator should document the date, time of the day and the reason for code breaking. If the code is broken, patient must discontinue IMP administration but continues the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diltiazem (Experimental): When signs of vascular dysfunction with the coronary function test.
  Interventions: Drug: Diltiazem Hydrochloride
- Placebo (Placebo Comparator): When signs of vascular dysfunction with the coronary function test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diltiazem Hydrochloride — Diltiazem hydrochloride is a calcium ion influx inhibitor (slow channel blocker or calcium antagonist). It is a white to off-white crystalline powder with a bitter taste. It is freely soluble in water, methanol and chloroform. It has a molecular weight of 450.98.
  It provides its therapeutic effects by blocking the influx of calcium ions into vascular smooth and cardiac muscle cells during membrane depolarization. The decrease in intracellular calcium causes relaxation of smooth muscle cells and cardiac myocytes by inhibiting actin-myosin interactions. Vasodilation subsequently results in decreased peripheral vascular resistance. The antihypertensive effect of diltiazem in hypertensives is greater than in normotensives.
  Diltiazem is registered for the treatment of hypertension, heart rate control in supraventricular tachycardia, chronic stable angina pectoris and angina pectoris resulting from coronary artery spasm.
  Other Names: Molecular Formula: C22H26N2S.HCl; Diltiazem HCl Retard 120 mg, Prolonged-Release Tablets; CAS 33286-22-5; Chemically diltiazem hydrochloride is the hydrochloride salt of (2S, 3S)-5-(2- Dimethylaminoethyl)- 2, 3, 4, 5-tetrahydro-2-(4-methoxyphenyl)-4-oxo-1, 5-benzothiazepin-3- yl-acetate
  Arms: Diltiazem
Drug: Placebo — Matching placebo capsules, given QD per oral use. Placebo capsules will be used in the same manner with the same dose titration.
  Arms: Placebo

SUMMARY:
Rationale: Up to 40% of patients undergoing a coronary angiogram for symptoms/signs of ischemia do not have obstructive coronary artery disease (CAD). In about half of them the mechanism underlying cardiac ischemia is coronary microvascular dysfunction (CMD). In CMD, myocardial ischemia is caused by impaired endothelial and/or non-endothelial coronary vasoreactivity resulting in the coronary microvasculature not dilating properly or becoming vasospastic. Recently published diagnostic criteria state that to confirm the diagnosis, CMD patients should either have an impaired coronary flow reserve (CFR), increased microvascular resistance (IMR) or have evidence of microvascular spasms. Hence, invasive coronary function testing (CFT) is considered the reference standard for a definitive diagnosis of CMD.

Patients with microvascular angina often have continuing episodes of chest pain leading to frequent first aid visits and hospital re-admissions with associated high health care costs. Moreover, CMD is associated with a worsened cardiovascular prognosis. Therefore, adequate treatment is paramount. However, current treatment options are based on a limited number of small studies, most of which were not placebo-controlled. Based on prior studies and our clinical experience we believe diltiazem, a calcium channel blocker (CCB) could improve coronary microvascular function in patients with CMD.

Objective: Our primary objective is to assess the effect of diltiazem on coronary microvascular function as assessed by CFT in symptomatic patients with CMD. Our secondary objective is to assess the effect of diltiazem on the individual coronary function parameters.

Study design: This is a clinical multi-center randomized with 1:1 ratio, double-blind, placebo-controlled study. Patients with chronic angina in the absence of obstructive CAD will be screened for study enrollment. Eligible patients will be asked for informed consent after which the screening visit will take place. Within 8 weeks after screening they will undergo CFT with the assessment of the coronary flow reserve (CFR), index of microcirculatory resistance (IMR) and coronary spasm.

* Intervention arm: if CFT shows either a CFR ≤ 2.0, an IMR ≥ 25 and/or coronary spasm, the patient will continue in the intervention arm of the trial and will be randomized to either diltiazem or placebo treatment for 6 weeks. After 6 weeks, a CFT will be repeated and the diltiazem/placebo treatment will be discontinued. Follow-up will be obtained after 6 weeks of treatment, and 1 year and 5 years after treatment discontinuation.
* Registration arm: If the CFT at baseline shows no signs of vascular dysfunction, patients will enter in the registration arm of the study. These patients will not receive any study medication. Follow-up will be obtained after 1 year and 5 years.

Study population: Adult patients with chronic angina in the absence of obstructive CAD will be screened for participation. They will be recruited from the outpatient clinic of the cardiology department of the participating sites. Patients with contra-indications for coronary function testing (with the use of adenosine and acetylcholine) and/or diltiazem treatment (i.e. severe AV conduction delay, hypersensitivity, reduced left ventricular function) will not be eligible.

Intervention: After establishing an abnormal coronary vascular function, 6 weeks treatment with either diltiazem 120-360 mg or placebo will be initiated in a double-blind fashion. Every two weeks dose titration will be performed if possible, under the guidance of patient tolerance (dizziness, leg oedema, etc.), blood pressure and heart rate.

Main study parameters/endpoints: The proportion of patients having a successful treatment with diltiazem, defined as normalization of at least one abnormal parameter and none of the normal parameters becoming abnormal.. A normal IMR is specified as IMR < 25, a normal CFR being a CFR > 2 and a normal acetylcholine test is specified as one without ECG abnormalities and without signs of spasm at the same acetylcholine dose used at baseline. Main secondary endpoints will be the change in the individual coronary function parameters.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The extensive experience with diltiazem and the favourable safety profile in combination with the short duration of treatment make the treatment risk low for participants. Related to the study procedure several reports show that CFT is a safe procedure with serious complication rates (death, myocardial infaction, etc.) ranging from 0 to 0.7%. The first CFT is clinically indicated by the treating physician. The second CFT will bring additive risk to the participants in the intervention arm. However, we believe it is essential to investigate the effect of diltiazem on coronary function to justify its use in CMD patients.

DETAILED DESCRIPTION:
Primary Objective:

To assess the effect of diltiazem on coronary microvascular function in patients with chronic angina and evidence of coronary microvascular dysfunction.

Secondary Objectives:

To assess the effect of 6 weeks of treatment with diltiazem on the individual coronary function parameters in patients with coronary microvascular dysfunction.

Safety objective:

To assess the safety of coronary function testing in patients with chronic angina in the absence of obstructive CAD.

To assess the safety of treatment with diltiazem in patients with coronary microvascular dysfunction.

Exploratory objectives:

To assess the effect of 6 weeks of treatment with diltiazem on angina frequency and severity in patients with coronary microvascular dysfunction.

To assess the difference in major adverse cardiovascular events (MACE) in symptomatic patients with and without coronary microvascular dysfunction at 1 and 5 year follow-up.

Sample size calculation:

There are little data available about the effect of oral diltiazem on coronary non-endothelium dependent and endothelium dependent vasoreactivity.

The effect of CCBs on non-endothelium dependent vasoreactivity: one randomized placebo-controlled study shows oral treatment with diltiazem improves TIMI frame count on repeat coronary angiography (1) In current practice, CFR and IMR quantitative measurements have replaced the TIMI frame count. Another non-placebo controlled study shows an improvement of echocardiography-measured CFR in CMD patients treated with 90mg diltiazem.(2) The effect of CCBs on endothelium dependent vasoreactivity: patients who are treated with ultra long-acting CCBs (i.e. amlodipine) show less vasoconstriction on baseline coronary angiography and have a lower rate of positive acetylcholine provocation testing compared to patients who don't (41% vs. 64%) if all of them stop all CCBs 48 hours before the procedure. (3) We find a 25% success rate of treatment with diltiazem clinically relevant. Based on the previous literature, that kind of treatment effect is expected to be feasible we anticipate a 30% success rate in the patients treated with diltiazem compared to a 5% success rate in those treated with placebo. To detect this difference with type I error rate of 5% and type II error rate of 80% we need a total of 72 subjects (36 in each group) in the study. Based on prior research, (2, 3) we estimate that at least 60% of the screened patients will have an abnormal coronary reactivity test. We estimate that 15% of the randomized patients will discontinue the IMP during the treatment phase due to side effects of diltiazem (gastro-intestinal side effects, peripheral oedema, see section 6.4) or inability to undergo the second coronary reactivity test. Therefore, a total of 142 patients needs to be screened to reach intended sample size of 72 patients that complete the study protocol, as shown in figure 2.

An interim analysis will be performed for futility when half of the patients has been recruited in both arms. The boundary for futility consideration will be a conditional power of <20% under the alternative hypothesis (4). At conditional power of <20% under original design effect assumption, a single assessment of futility when half of the patients has been recruited in both arms, we expect very limited inflation in type II error rate. (5, 6)

Statistical analysis:

For summarizing patient characteristics, continuous variables with a Gaussian distribution will be expressed as mean ± standard deviation (SD), and continuous variables with a non-Gaussian distribution as median ± interquartile range (IQR). Categorical variables will be summarized with number (percentage).

Analysis Populations:

The full analysis population will consist of all patients who signed informed consent from both the intervention arm and the registration arm.

All patients who are enrolled in the intervention arm of the study and are randomly allocated to treatment or placebo group will be included in the primary analysis of efficacy (intention-to-treat treat analysis, ITT).

In a supportive analysis, the Per Protocol (PP) group will consist of all patients from the ITT group without major protocol violations. Major protocol violations are:

* In- or exclusion criteria are not met
* Inadequate informed consent
* Serious non-compliance of the IMP: a drug-compliance < 80%
* Missing data: subject who misses primary outcome data from the first and/or second CFT (acetylcholine testing outcome, CFR and IMR data).

The safety population will be the as-treated population, which will consist of all patients from the intervention group who had at least one dose of trial medication.

Data Safety Monitoring Board (DSMB):

A DSMB will be formed for two analyses: one interim look after half of the patients (as calculated in the original power analysis) completed visit 104 (the second coronary reactivity test), and one analysis after all 72 patients completed visit 104. The full procedure is described in the DSMB Charter.

The DSMB would be responsible for the execution of the interim analysis and for making recommendations to the executive committee based on a clearly defined written charter. The objective of the interim analysis will be to assess the following:

* Safety issue: is there any difference in the safety profile between treatment groups? If yes, are these associated with drug administration?
* Futility: is it unlikely that a relevant treatment difference will be demonstrated?
* Efficacy: do the data show an overt efficacy of diltiazem compared to placebo?
* Are there any other observations in the accumulated data that should be communicated to the sponsor? The advice(s) of the DSMB will be sent to the sponsor of the study. Should the sponsor decide not to fully implement the advice of the DSMB, the sponsor will send the advice to the reviewing METC, including a note to substantiate why (part of) the advice of the DSMB will not be followed.

Regulation statement:

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/GCP and in accordance with the Medical Research Involving Human Subjects Act (WMO) and other guidelines, regulations and Acts

Recruitment and consent:

The Principal Investigator(s) will:

* Ensure each patient is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study.
* Ensure each patient is notified that they are free to discontinue from the study at any time.
* Ensure that each patient is given the opportunity to ask questions and allowed time to consider the information provided.
* Ensure each patient provides signed and dated informed consent before conducting any procedure specifically for the study.
* Ensure the original, signed Informed Consent Form(s) is/are stored in the Investigator's Study File.
* Ensure a copy of the signed Informed Consent Form is given to the patient.
* Ensure that any incentives for patients who participate in the study as well as any provisions for patients harmed as a consequence of study participation are described in the informed consent form that is approved by an Ethics Committee.

Patients with angina in the absence of obstructive CAD will be screened for participation in the study according to the the Inclusion criteria and Exclusion criteria. Most of these patients will be identified from the waiting list for a CFT. Patients will only be eligible if the treating physician has already agreed with the patient to perform a CFT for his/her angina. After the patient has agreed to be informed about the study he/she will be contacted by one of the members of the study team and will receive the patient information. Preferably, a face-to-face information visit will be planned 1-2 weeks after the patient information was provided (but before the coronary reactivity test). The alternative would be a telephone visit to explain the patient information. Only after the patient is well informed, all questions are answered and he/she agrees to participate, the screening visit will be planned where the informed consent form will be signed. If the patient does not want to participate in the study, the coronary reactivity test will still take place.

Benefits and risks assessment, group relatedness:

It is essential to only include patients with properly diagnosed CMD patients without current obstructive CAD and an abnormal coronary reactivity. To assess both endothelial-dependent and endothelial-independent coronary vasoreactivity, invasive CFT is currently the only diagnostic option.

Wei et al., report on the safety of invasive CFT in women to diagnose CMD.(7) Among 293 symptomatic women without obstructive CAD who underwent testing, four total adverse events occurred - two of which were deemed serious: a coronary dissection and an episode of coronary spasm leading to acute myocardial infarction. Over the course of > 5 year follow-up, the overall rate of major adverse cardiac events in the population was 8.2%. The investigators rightly conclude that the immediate risk of testing is relatively low in comparison to the overall event rate in this population. Ong et al. also report low risk of coronary function testing using ACH testing in 124 patients without obstructive CAD.(28) There were no serious complications (e.g., myocardial infarction, refractory spasm, sustained ventricular arrhythmias, or need for resuscitation). Transient atrioventricular block was frequently observed and occurred mostly during provocation of the RCA; it always resolved within seconds after reducing the speed of the ACH injection, due to the short half-life of ACH. We will not include testing of the RCA in our protocol.

In our clinical experience, diltiazem relieves angina in patients with CMD. To justify the use of this agent in the treatment of CMD it is essential to prove its effect on coronary reactivity (besides its effect on symptoms). Diltiazem is widely used, cheap and safe. Its characteristics are promising with regard to it's potential to improve coronary vasoreactivity.

Handling and storage of data and documents:

The data generated will be encoded and a separate patient identification log will be created. The key to the code will only be available to the principal investigator and delegated investigators. The acquired encoded data imputed in the eCRF will be accessible with passwords to the researchers involved. Personal data will comply to the Dutch Personal Data Protection Act.

Monitoring and Quality Assurance:

During the study, the study sites will be monitored to review study progress, Investigator and patient compliance with clinical protocol requirements and any emergent problems. The monitor visit will include: patient informed consent, patient recruitment and follow-up, SAE documentation and reporting, AE documentation, IMP allocation, IMP accountability and quality of the data. Details will be specified in a monitoring plan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic angina, defined as symptoms of angina at least 2 times a week despite medical therapy for the last 3 months.
* No signs of obstructive coronary artery disease (CAD), documented within 5 years* before inclusion by one of the following modalities:

  * Patients with non-obstructive (< 50% stenosis) coronary arteries, or patients with one or more intermediate stenoses (between 50 and 70%) with documented FFR > 0.80 or iFR > 0.89 on angiogram.
  * Coronary computed tomography angiography (CCTA) with finding of non-obstructive coronary arteries
* Baseline coronary function testing with at least one of the following:

  1. CFR ≤ 2.0
  2. IMR ≥ 25
  3. Abnormal acetylcholine test defined as the presence of (recognizable) angina, ischemic ECG abnormalities with or without epicardial spasm.
* Signed written informed consent * Note: in cases of clinically suspected progression of atherosclerosis as per the Investigator, more contemporary (i.e., 6 months) evidence should be provided.

Exclusion Criteria:

* Other cause of angina deemed highly likely by the treating physician.
* Active use of calcium channel blockers or any use of calcium channel blockers in the previous two weeks or known intolerance for non-dihydropyridine calcium channel blockers.
* Left ventricular ejection fraction < 50%.
* Recent PCI within the past 3 months.
* Patients with history of coronary artery bypass grafting (CABG).
* Surgically uncorrected significant congenital or valvular heart disease, cardiomyopathy or myocarditis.
* Significant renal impairment (eGFR < 30).
* Significant hepatic impairment (history or cirrhosis or abnormal serum ALT or AST 3-fold greater than the upper limit of normal).
* Pregnant women or women of child bearing potential who are planning to become pregnant within the next 3 months.
* Prior non-cardiac illness with an estimated life expectancy < 1 year.
* Contra-indication to coronary function testing:

  1. Contraindication or known hypersensitivity to adenosine.
  2. Contraindication or known hypersensitivity to acetylcholine.
  3. Ongoing dipyridamole treatment.
* Contra-indication for treatment with CCB: second or third degree AV block, sinus node dysfunction, bradycardia (heart rate < 50 beats/minute) and/or potentially dangerous interaction due to the use of another CYP3A4 substrate in the opinion of the investigator.
* Symptomatic hypotension or systolic BP < 100 mmHg at screening visit on 2 consecutive measurements.
* History of hospitalization for asthma and/or current use of ≥ 2 types of pulmonary medications for asthma and/or severe COPD with FEV1 < 50% of predicted.
* Participation in another clinical study with an IMP within one month prior to enrolment.
* Inability of the patient, in the opinion of the investigator, to understand and/or comply with study medications, procedures and/or follow-up OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study.
* Unable to give informed consent (i.e. due to language barrier).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients having a successful treatment with diltiazem, defined as normalization of at least one abnormal parameter and none of the normal parameters becoming abnormal. | 6 weeks
  A normal IMR is specified as IMR < 25, a normal CFR being a CFR > 2 and a normal acetylcholine test is specified as one without spasm, without ischemic ECG abnormalities and without (recognizable) angina at the same acetylcholine dose used at baseline.

SECONDARY OUTCOMES:
Change in index of microvascular resistance (IMR) | 6 weeks
  the delta between 1st and 2nd coronary function test
Change in Coronary Flow Reserve (CFR) | 6 weeks
  the delta between 1st and 2nd coronary function test
Change in Acetylcholine test parameters | 6 weeks
  his is defined as the difference between the dose of acetylcholine at which the baseline CFT showed signs of spasm, compared to the dose at the second CFT. This will be compared between treatment and placebo group using a multinominal logistic regression. The efficacy population will be used for this analysis.
Change in Absolute flow parameters - flow (Q) (ml/min) | 6 weeks
  These are derived by subtracting the outcome from the second CFT from the outcome of the first CFT. To compare change in CFT parameters between treatment and placebo group, we will use independent sample t-test. Bonferroni correction will be applied to account for multiple testing. The efficacy population will be used for this analysis.
Change in Absolute flow parameters - Resistance (R) | 6 weeks
  These are derived by subtracting the outcome from the second CFT from the outcome of the first CFT. To compare change in CFT parameters between treatment and placebo group, we will use independent sample t-test. Bonferroni correction will be applied to account for multiple testing. The efficacy population will be used for this analysis.

OTHER OUTCOMES:
Safety endpoints | 6 weeks
  The occurrence of complications related to the coronary angiography and/or CFT will be collected, as well as adverse events related to the IMP.
Follow-up (MACE) | 5 years
  Number of major adverse cardiovascular events (MACE) at 1 and 5 year follow-up. MACE is defined as nonfatal stroke, nonfatal myocardial infarction, cardiovascular death, all-cause death, hospitalization for heart failure.
Change in angina frequency reporting in the patient diary | 5 years
  Change in patient reported outcome measures (PROs). These are derived by subtracting the outcome from the PROs from visit 104 to those from visit 1. The efficacy population will be used for this analysis.To compare change in PROs between treatment and placebo group, we will use independent sample t-test.
Change in the Seattle Angina Questionnaire (SAQ) | 5 years
  Change in patient reported outcome measures (PROs). These are derived by subtracting the outcome from the PROs from visit 104 to those from visit 1. The efficacy population will be used for this analysis.To compare change in PROs between treatment and placebo group, we will use independent sample t-test.
Change in RAND-36 scores | 5 years
  Change in patient reported outcome measures (PROs). These are derived by subtracting the outcome from the PROs from visit 104 to those from visit 1. The efficacy population will be used for this analysis.To compare change in PROs between treatment and placebo group, we will use independent sample t-test.
Change in angina CCS classification | 5 years
  Change in patient reported outcome measures (PROs). These are derived by subtracting the outcome from the PROs from visit 104 to those from visit 1. The efficacy population will be used for this analysis.To compare change in PROs between treatment and placebo group, we will use independent sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Elias-Smale, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Catharina Hospital, Eindhoven
  - Maasstad Hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li L, Gu Y, Liu T, Bai Y, Hou L, Cheng Z, Hu L, Gao B. A randomized, single-center double-blinded trial on the effects of diltiazem sustained-release capsules in patients with coronary slow flow phenomenon at 6-month follow-up. PLoS One. 2012;7(6):e38851. doi: 10.1371/journal.pone.0038851. Epub 2012 Jun 27. PMID 22761709
- [Background] Zhang X, Li Q, Zhao J, Li X, Sun X, Yang H, Wu Z, Yang J. Effects of combination of statin and calcium channel blocker in patients with cardiac syndrome X. Coron Artery Dis. 2014 Jan;25(1):40-4. doi: 10.1097/MCA.0000000000000054. PMID 24256699
- [Background] Kurabayashi M, Asano M, Shimura T, Suzuki H, Aoyagi H, Yamauchi Y, Okishige K, Ashikaga T, Isobe M. Ultra-long acting calcium channel blockers may decrease accuracy of the acetylcholine provocation test. Int J Cardiol. 2017 Jun 1;236:71-75. doi: 10.1016/j.ijcard.2017.02.123. Epub 2017 Feb 28. PMID 28268085
- [Background] Yeatts SD, Martin RH, Coffey CS, Lyden PD, Foster LD, Woolson RF, Broderick JP, Di Tullio MR, Jungreis CA, Palesch YY; IMS III Investigators. Challenges of decision making regarding futility in a randomized trial: the Interventional Management of Stroke III experience. Stroke. 2014 May;45(5):1408-14. doi: 10.1161/STROKEAHA.113.003925. Epub 2014 Apr 3. PMID 24699059
- [Background] Lachin JM. A review of methods for futility stopping based on conditional power. Stat Med. 2005 Sep 30;24(18):2747-64. doi: 10.1002/sim.2151. PMID 16134130
- [Derived] Jansen TPJ, de Vos A, Elias-Smale SE, Paradies V, Konst RE, Crooijmans C, Dimitriu-Leen AC, Rodwell L, Maas AHEM, Smits PC, van Royen N, Damman P. Effect of Diltiazem Versus Placebo on Microvascular Dysfunction Assessed By Repeated Continuous Thermodilution Measurements: Results of the EDIT-CMD Trial. J Am Heart Assoc. 2023 Nov 7;12(21):e030188. doi: 10.1161/JAHA.123.030188. Epub 2023 Oct 27. No abstract available. PMID 37889203
- [Derived] Jansen TPJ, Konst RE, de Vos A, Paradies V, Teerenstra S, van den Oord SCH, Dimitriu-Leen A, Maas AHEM, Smits PC, Damman P, van Royen N, Elias-Smale SE. Efficacy of Diltiazem to Improve Coronary Vasomotor Dysfunction in ANOCA: The EDIT-CMD Randomized Clinical Trial. JACC Cardiovasc Imaging. 2022 Aug;15(8):1473-1484. doi: 10.1016/j.jcmg.2022.03.012. Epub 2022 Apr 2. PMID 35466050